CLINICAL TRIAL: NCT01302756
Title: The Effect of High Dose Folic Acid Versus Placebo on the Rate of Gestational Diabetes or Gestational Hypertension in Pregnant Women: a Randomized Controlled Trial.
Brief Title: The Effect of High Dose Folic Acid Versus Placebo on the Rate of Gestational Diabetes or Gestational Hypertension in Pregnant Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: FWH20110006H
Record Dates: First submitted 2011-02-17; First posted 2011-02-24 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Gestational Diabetes; Gestational Hypertension
Keywords: gestational diabetes; gestational hypertension; folic acid
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Placebo — Group 1: Placebo plus standard of care pre-natal vitamins (which include 1 milligram of folic acid) a day for the duration of pregnancy
Dietary Supplement: Folic Acid — Group 2: 4-milligrams of folic acid a day for the duration of pregnancy plus standard of care pre-natal vitamins (which include 1 milligram of folic acid)

SUMMARY:
The purpose of this study is to determine if higher-than usual doses of daily folic acid has an effect on the rate of gestational diabetes mellitus (GDM) or gestational hypertension in pregnant women while determining status of folic acid, vitamin B12, homocysteine and vitamin D in pregnancy.

DETAILED DESCRIPTION:
Subjects (DoD beneficiaries) will be recruited from all non-diabetic female subjects whom are at least 18 years of age and are empanelled for care at Nellis Air Force Base. Upon arrival at the mandatory New Obstetrics (OB) Orientation, potential subjects will be offered an opportunity to participate in this study. A total of 650 subjects will be recruited. After consent and HIPAA Authorization is obtained, the subjects will have Baseline blood pressure, fasting glucose, folic acid, vitamin B12, homocysteine, vitamin D measurements, and weight, height, race, ethnicity, parity, vegetarian status recorded. Subjects will be written a prescription and sent to the Clinical Pharmacy where they will be randomized via block randomization. After randomization, they will receive either placebo or 4 milligrams of folic acid (in addition to the standard of care pre-natal vitamins) from the pharmacy--thus investigators and subjects will be blinded as to their treatment.

Group 1: Placebo plus standard of care pre-natal vitamins (which include 1 milligram of folic acid) a day for the duration of pregnancy Group 2: Will take an additional 4-milligrams of folic acid a day for the duration of pregnancy plus standard of care pre-natal vitamins (which include 1 milligram of folic acid)

The Placebo will be a gelatin capsule filled with starch which does not increase the risks to subjects.

The pre-natal vitamins dispensed at the MOFH Clinical Pharmacy include 1 milligram of folic acid. The folic acid is manufactured by West Ward Pharmaceutical Corp.

Those subjects in Group 2 will be taking a total of 5 milligrams of folic acid (1 milligram of folic acid is contained in their standard of care pre-natal vitamins and they will be given an additional 4 milligrams of folic acid as part of this research study).

The placebo is manufactured by Green Valley Medical Supply Company.

Subjects will continue to receive routine obstetrics care and take their prescription for the duration of their pregnancy. Per the American College of Obstetrics and Gynecology (ACOG), patients will be tested for gestational diabetes either at 2nd trimester for those with risk factors of prior GDM, age >34 or body mass index >25 or at 28 weeks for standard risk women. There will be an unblinded person to monitor any adverse effects that may occur.

At 28 weeks gestation, weight, height, diagnosis of GDM, gestational hypertension, pre-eclampsia, post-partum hemorrhage, maternal death will be recorded, and will be asked if they took the study medications as prescribed (studies have shown that patient recall is as accurate as pill counts).

At delivery, folic acid, B12, homocysteine, vitamin D will be measured and weight, height, diagnosis of GDM, gestational hypertension, pre-eclampsia, post-partum hemorrhage, maternal death, birth weight, shoulder dystocia, neonatal/fetal mortality will be recorded, and will be asked if they took the study medications as prescribed (studies have shown that patient recall is as accurate as pill counts).

After completion of the first 200 subjects, an interim power analysis to identify whether the trial can be stopped early. At this point and at the conclusion of the study, the data will be de-identified and analyzed. A paper will be written and submitted to a scientific journal at the conclusion of the study.

When subjects have completed the study, the Pharmacy will then de-randomize the information and send to the Principal Investigator for analysis.

If at any time during the study, the subject decides to withdraw from the study, they will be referred to their Primary Care Manager to initiate standard of care treatment.

If any subjects experience fetal demise or maternal death, the Principal Investigator will consult with Obstetrics to initiate proper clinical care.

Folic acid is a common supplement in pregnancy.

"In accordance with 21 CFR 312.2(b)(i-v), an IND exemption is requested based on the following provisions: (i) The investigation is not intended to be reported to FDA as a well-controlled study in support of a new indication for use nor intended to be used to support any other significant change in the labeling for the drug; (ii) If the drug that is undergoing investigation is lawfully marketed as a prescription drug product, the investigation is not intended to support a significant change in the advertising for the product; (iii) The investigation does not involve a route of administration or dosage level or use in a patient population or other factor that significantly increases the risks (or decreases the acceptability of the risks) associated with the use of the drug product; (iv) The investigation is conducted in compliance with the requirements for institutional review set forth in part 56 and with the requirements for informed consent set forth in part 50; and (v) The investigation is conducted in compliance with the requirements of §312.7."

ELIGIBILITY:
Inclusion Criteria:

* Tricare Insurance Beneficiary (military insurance) receiving care at Nellis AFB
* Pregnant females (DoD beneficiaries) at least 18 years of age

Exclusion Criteria:

* Diagnosed as being diabetic
* Diagnosed with chronic hypertension prior to pregnancy
* Personal or family history of neural tube defects or personal history of birth defects
* Unable to communicate
* Non-English speaking
* Patients who know they will move prior to delivery
* Patients who have had Gastric Bypass surgery
* Patients with known seizure disorder or on anti-seizure medication
* Patients taking a folic acid antagonist
* Patients who are hypohomocysteine
* Previously diagnosed with Methylenetetrahydrofolate reductase (MTHFR) mutation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes | 2 years
  Subjects will have baseline blood levels drawn for fasting glucose, folic acid, vitamin B12, homocysteine and vitamin D measurements. They will be randomized to take either standard of care dose of folic acid or an additional 4 milligrams of folic acid for the duration of their pregnancy. The blood levels will again be drawn for fasting glucose, folic acid, vitamin B12, homocysteine and vitamin D measurements.

SECONDARY OUTCOMES:
Gestational hypertension | 2 years
  Subjects will have baseline blood levels drawn for fasting glucose, folic acid, vitamin B12, homocysteine and vitamin D measurements. They will be randomized to take either standard of care dose of folic acid or an additional 4 milligrams of folic acid for the duration of their pregnancy. The blood levels will again be drawn for fasting glucose, folic acid, vitamin B12, homocysteine and vitamin D measurements.